CLINICAL TRIAL: NCT03067350
Title: Influence of a Combined Pharmacogenetic Score on Through Plasma Voriconazole Concentrations in Haematological Patients
Acronym: VORIGENE
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC15.168
Record Dates: First submitted 2017-02-06; First posted 2017-03-01 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Invasive Aspergillosis; Haematological Cancer Patients; Voriconazole
Keywords: voriconazole; pharmacogenetics; pharmacokinetics; therapeutic drug monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hypothesis: A pharmacogenetic score integrating both CYP3A genotypes could be influence initial trough voriconazole plasma concentrations and thus useful to adapt a priori voriconazole dosing in order to get adequate voriconazole exposure as possible after starting treatment.

Main Objective: To determine predictive value of a combined pharmacogenetic score on onset of trough voriconazole plasma concentration inferior than lower therapeutic target.

DETAILED DESCRIPTION:
Voriconazole (VRC), the gold-standard treatment of invasive aspergillosis is characterized by variables and nonlinear pharmacokinetics, causing many under- or over-dosing. A link exist between trough plasma concentrations (Cmin) of VRC and effectiveness but also its toxicity. Thus the longitudinal therapeutic drug monitoring of VRC is now recommended with a therapeutic range between 1 and 5 mg/L. The pharmacokinetic variability of VRC is in part explained by its metabolism, mainly dependent on cytochrome P 450 (CYP), particularly CYP2C19, 3A4, 3A5; all these CYP exhibiting genetic polymorphisms. The authors, recently shown, and for the first time , in a retrospective study conducted in 29 patients allogeneic hematopoietic stem cell that initial VRC Cmin adjusted the dose was not only influenced by the route of administration but also by a pharmacogenetics score whose determination is to assign each genotype CYP2C19 and CYP3A a score expressed in a arbitrary units.

The combined pharmacogenetic score was strongly correlated with the original Cmin (r= -0.748; p = 0.002) and was the only independent predictor of initial Cmin (after adjusting the dose and the route of administration). In addition, none of the patients having a genetic score <2 (ie metabolizing capacity of reduced VRC) did not show an initial Cmin below 1 mg/L, while the initial Cmin was below this threshold efficiency in 47% of patients with a genetic score >2. The aim of this new study is to confirm the impact of the pharmacogenetic score on the initial VRC Cmin over a larger prospective cohort of 60 adult patients with onco-hematological diseases.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from haematological cancer

Exclusion Criteria:

* less than 18-years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients suffering from haematological cancer Followed at the hematolofic clinic of Grenoble University Hospital Starting treatment by voriconazole whatever the route of administration
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
number of initial voriconazole trough plasma concentration in the therapeutic range (1-4mg/l) | concentration measured between 5 to 10 days after voriconazole treatment initiation
  Initial voriconazole trough plasma concentration

SECONDARY OUTCOMES:
initial voriconazole trough plasma concentrations adjusted on the dose | concentration measured between 5 to 10 days after voriconazole treatment initiation
  Initial voriconazole trough plasma concentration
number of patients with therapeutic success | 3 months after voriconazole therapy initiation
  treatment outcome determined 3 months after voriconazole initiation (failure, stable response, success)
number of patients with adverse effects | duration of voriconazole treatment (maximum length of follow-up : 3 months)
  adverse effects include neurological disorders such as visual disturbance and/or hallucinations and hepatotoxicity (evaluated by ALAT/ASAT, bilirubin and γ-GT levels),

CONTACTS AND LOCATIONS:
Overall Officials: Elodie GAUTIER, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital, Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gautier-Veyret E, Fonrose X, Tonini J, Thiebaut-Bertrand A, Bartoli M, Quesada JL, Bulabois CE, Cahn JY, Stanke-Labesque F. Variability of voriconazole plasma concentrations after allogeneic hematopoietic stem cell transplantation: impact of cytochrome p450 polymorphisms and comedications on initial and subsequent trough levels. Antimicrob Agents Chemother. 2015 Apr;59(4):2305-14. doi: 10.1128/AAC.04838-14. Epub 2015 Feb 2. PMID 25645831
- [Background] Gautier-Veyret E, Fonrose X, Stanke-Labesque F. A genetic score combining CYP450 2C19 and 3A4 genotypes to predict voriconazole plasma exposure? Int J Antimicrob Agents. 2016 Aug;48(2):221-2. doi: 10.1016/j.ijantimicag.2016.05.002. Epub 2016 Jun 7. No abstract available. PMID 27318623
- [Background] Tonini J, Bailly S, Gautier-Veyret E, Wambergue C, Pelloux H, Thiebaut-Bertrand A, Cornet M, Stanke-Labesque F, Maubon D. Contribution of a Simple Bioassay in Effective Therapeutic Drug Monitoring of Posaconazole and Voriconazole. Ther Drug Monit. 2015 Oct;37(5):685-8. doi: 10.1097/FTD.0000000000000199. PMID 26384041
- [Background] Tonini J, Thiebaut A, Jourdil JF, Berruyer AS, Bulabois CE, Cahn JY, Stanke-Labesque F. Therapeutic drug monitoring of posaconazole in allogeneic hematopoietic stem cell transplantation patients who develop gastrointestinal graft-versus-host disease. Antimicrob Agents Chemother. 2012 Oct;56(10):5247-52. doi: 10.1128/AAC.00815-12. Epub 2012 Jul 30. PMID 22850515
- [Background] Jourdil JF, Tonini J, Stanke-Labesque F. Simultaneous quantitation of azole antifungals, antibiotics, imatinib, and raltegravir in human plasma by two-dimensional high-performance liquid chromatography-tandem mass spectrometry. J Chromatogr B Analyt Technol Biomed Life Sci. 2013 Mar 1;919-920:1-9. doi: 10.1016/j.jchromb.2012.12.028. Epub 2013 Jan 9. PMID 23384531